CLINICAL TRIAL: NCT07376265
Title: Comparative Effectiveness of Sacubitril/Valsartan vs ACEi/ARB in HFrEF Patients: Real Heart PT
Brief Title: A Real-world Study to Compare the Effectiveness of Sacubitril/Valsartan Versus ACEi/ARB in HFrEF Patients
Status: Completed | Type: Observational
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Other Study IDs: CLCZ696BPT07
Record Dates: First submitted 2026-01-22; First posted 2026-01-29 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-01

CONDITIONS: Heart Failure
Keywords: Sacubritril-valsartan; Heart failure; Cardiovascular outcomes
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (3):
- SAC/VAL Cohort: Adult patients with HFrEF undergoing therapy with SAC/VAL.
- ACEi/ARB Cohort: Adult patients with HFrEF undergoing therapy with ACEi/ARB.
- Missed Opportunities Cohort: Patients who were eligible for but did not receive SAC/VAL.

SUMMARY:
This was a retrospective, observational, comparative cohort study using secondary data from electronic health records (EHR) from a local health unit that provides primary, secondary and tertiary care to a resident population in northern Portugal. The study aimed to assess the comparative effectiveness of sacubitril/valsartan (SAC/VAL) versus angiotensin-converting enzyme inhibitors (ACEi) or angiotensin receptor blockers (ARB) in patients with heart failure with reduced ejection fraction (HFrEF).

ELIGIBILITY:
Inclusion criteria:

* Left ventricular ejection fraction (LVEF) < 40%
* Brain natriuretic peptide (BNP) ≥35 pg/mL or N-terminal prohormone of brain natriuretic peptide (NT-proBNP) ≥125 pg/mL
* Had a record in the database in the 365 days prior to the index date

Exclusion criteria:

* Missing sex or date of birth
* Estimated glomerular filtration rate (eGFR) below 30 mL/min/1.73 m^2 at SAC/VAL, ACEi or ARB initiation
* History of angioedema or unacceptable side effects during receipt of SAC/VAL, ACEi or ARB
* Severe hepatic impairment, biliary cirrhosis, and cholestasis
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study included heart failure patients with reduced ejection fraction.
Sampling Method: Non-Probability Sample
Enrollment: 1249 (Actual)
Dates: Start 2023-10-20 (Actual); Primary Completion 2024-04-11 (Actual); Study Completion 2024-04-11 (Actual)

PRIMARY OUTCOMES:
Hazard Ratio for the Composite of Cardiovascular Death or Heart Failure Hospitalization | 180 days, 810 days, 1260 days

SECONDARY OUTCOMES:
Hazard Ratio for Death From Cardiovascular Causes | 180 days, 810 days, 1260 days
Hazard Ratio for Hospitalization for Heart Failure | 180 days, 810 days, 1260 days
Hazard Ratio for First Hospitalization or Emergency Room Visit | 180 days, 810 days, 1260 days
  Hospitalizations or emergency room visits for heart failure, and any cause were recorded.
Hazard Ratio for First Cardiovascular-specific Hospitalization | 180 days, 810 days, 1260 days
Hazard Ratio for the Composite of Death From Cardiovascular Causes, Hospitalization for Heart Failure, Non-fatal Myocardial Infarction and Non-fatal Stroke | 180 days, 810 days, 1260 days
Hazard Ratio for Implantable Cardioverter-defibrillator (ICD) Procedure | 180 days, 810 days, 1260 days
Hazard Ratio for All-cause Mortality | 180 days, 810 days, 1260 days
Hazard Ratio for Improved LVEF | 180 days, 810 days, 1260 days
  Improved LVEF was defined as having at least one LVEF measurement equal or above 40% after having an LVEF under 40%.
Pearson Correlation Coefficient Between Change From Baseline in NT-proBNP and LVEF | 180 days, 810 days, 1260 days
Change From Baseline in NT-proBNP | 180 days, 810 days, 1260 days
Change From Baseline in LVEF | 180 days, 810 days, 1260 days
Total Healthcare Resource Utilization Costs per Calendar Year | Up to 5 years
  Healthcare utilization costs included costs for inpatient care, outpatient care, medication, and exams.
Number of Days Patients Were Absent From Work per Calendar Year | Up to 5 years
Healthcare Resource Utilization Costs per Patient per Year | Up to 5 years
  Healthcare utilization costs included costs for inpatient care, outpatient care, medication, and exams.
Hazard Ratio for Hyperkalemia | 180 days, 810 days, 1260 days
Rate of Dose Titration Events per 100-Person-Years | 180 days, 810 days, 1260 days
  Rates were measured for dose titrations from:
  * low to medium
  * medium to low
  * medium to high
  * high to medium
Rate of Patients Reaching the Maximum Dose per 100-Person-Years | 180 days, 810 days, 1260 days
Rate of Treatment Discontinuation | 180 days, 810 days, 1260 days
Number of Patients by Demographic Category | Baseline
  Demographics included age and sex.
Number of Patients by Clinical Characteristic Category | Baseline
  Clinical characteristics included:
  * New York Heart Association (NYHA) Class
  * eGFR ≥ 60 mL/minute/1.73 m^2
  * eGFR < 60 mL/minute/1.73 m^2
  * LVEF ≤ 35%
  * LVEF > 35%
  * Type of medication
  * Comorbidities

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (1):
- Novartis, East Hanover, New Jersey, United States

REFERENCES:
- See also: Link to study results — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=18409